CLINICAL TRIAL: NCT02805413
Title: Simultaneous Determination of Blood Pressure by Oscillometry and Photoplethysmography Compared to the Standard Inert Gas Rebreathing Technique
Acronym: CeCi
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Collaborators: Novespace (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2015-A00264-45
Record Dates: First submitted 2016-04-21; First posted 2016-06-20 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: BLOOD PRESSURE

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DETERMINATION OF BLOOD PRESSURE (Other): determination and comparison of blood pressure by/with :
  * Pulse Curve Analysis
  * Inert gas re-breathing
  * Central blood pressure device
  * Vascular ultrasound device
  * Thoracic Impedance (ICG) - Electrocardiography (ECG) - Phonocardiography (Phono) - Carotid plethysmography (Pneumo)
  Interventions: Other: Détermination and comparison of blood pressure

INTERVENTIONS:
Other: Détermination and comparison of blood pressure — Rebreathings will be performed every parabola (2, 4, 6, 8, 10…). Ultrasound measurements will be performed during the remaining parabolas (1, 3, 5, 7, 9…). The procedure consists of a fixed breathing frequency of 20 breaths per minute and an exact triggered start point for the measurements. . Central blood pressure measurements, finger blood pressure measurements, impedance cardiography, carotid plethysmography and phonocardiography will be performed continuously during the flights. The breaks between parabolas 10 and 11 and 20 and 21 will be used to change subjects, which takes approximately 5 minutes.

SUMMARY:
Main objective of the experiment is threefold: 1) to technically test a device for central blood pressure estimation for its applicability in a spaceflight-related environment and on the International Space Station. 2) Furthermore the objective is to compare central blood pressure estimates based on arterial pressure readings of different peripheral arteries. For central blood pressure estimation mathematical transfer functions as described by Karamanoglu and colleagues (11) will be used. 3) Finally the experiments' objective is to simultaneously apply phonocardiography together with ECG and carotid plethysmography to determine cardiac systolic time intervals in parabolic flight during gravity transitions.

Secondary objective of the experiment is to simultaneously measure key variables of the central circulation during gravity transitions to expand the understanding of cardiovascular regulation in weightlessness. Furthermore spirometric measurements shall be performed during a parabolic flight day to observe changes in end-expiratory CO2. Arterial CO2 content is central for cardiovascular regulation.

Our main hypothesis is that there is no difference between different methods of central arteria pressure determination.

Concerning our secondary objective, this experiment is designed as an observational study. Thus no clear hypothesis was generated but the measured cardiovascular and respiratory variables will be analysed regarding differences correlated to gravity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (men or women)
* Aged from 18 to 65
* Affiliated to a Social Security system and, for non-French resident, holding a European Health Insurance Card (EHIC)
* Who accepted to take part in the study
* Who have given their written stated consent
* Who has passed a medical examination similar to a standard aviation medical examination for private pilot aptitude (JAR FCL3 Class 2 medical examination). There will be no additional test performed for subject selection.

Subjects will be staff member of the team or of other teams participating in the parabolic flight campaign

Exclusion Criteria:

* Person who took part in a previous biomedical research protocol, of which exclusion period is not terminated
* Treated or non-treated arterial hypertension
* Pregnant women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2015-04; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Central arterial pressure | baseline and when in gravity (same day)
  Central arterial pressure evaluated by oscillographic upper arm measurements

SECONDARY OUTCOMES:
Systolic time intervals | baseline and when in gravity (same day)
  Systolic time intervals evaluated in upright subjects regarding g-load.
inert gas rebreathing | baseline and when in gravity (same day)
  Cardiac output by inert gas rebreathing
heart rate | baseline and when in gravity (same day)
peripheral blood pressure | baseline and when in gravity (same day)
different methods of pulse curve analysis | baseline and when in gravity (same day)
  Cardiac output by different methods of pulse curve analysis will be evaluated for different g-loads.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre DP Denise, PhD, Principal Investigator — CHU CAEN
Locations (1):
- Caen CHU, Caen, France

IPD SHARING:
Plan to Share IPD: No